CLINICAL TRIAL: NCT04720755
Title: Low Intensity Extracorporeal Shock Wave Therapy (Li-ESWT) for Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1572819
Record Dates: First submitted 2020-12-15; First posted 2021-01-22 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction; Low intensity shock wave therapy
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Participants will receive twice-weekly Li-ESWT treatments of 0.2mJ/mm² over 3 treatment sites along the dorsal penile shaft (distal, mid-shaft, proximal), 1500 shocks per treatment (500 shocks per treatment site) for a total of 3000 shocks per week, for 6 weeks (total of 18,000 shocks)
  Interventions: Device: Low-Intensity Extracorporeal Shock Wave Therapy

INTERVENTIONS:
Device: Low-Intensity Extracorporeal Shock Wave Therapy — Twice-weekly treatments for 6 weeks, of 0.2mL/mm^2 administered for 500 shocks per treatment site, for a total of 3000 shocks per week.
  Other Names: Storz Duolith SD-1 t-top >>ultra<< device

SUMMARY:
Low-intensity extracorporeal shock wave therapy (Li-ESWT) has shown promise as a novel treatment for erectile dysfunction (ED), though the the mechanism of action and optimal protocol for administration has not been well-established. The aim of this study is to assess for subjective and objective improvements in erectile function following treatment with Li-ESWT.

DETAILED DESCRIPTION:
Eligible patients will be enrolled as outlined below. Prior to initiation of Li-ESWT treatments, patients will complete validated questionnaires to assess erectile function. In addition, patients will undergo induction of artificial erection in clinic with assessment of penile blood flow using penile Doppler. Intracavernosal pressure measurements will be obtained. A corporal aspirate will be drawn and examined for levels of neuronal nitric oxide synthase, endothelial nitric oxide synthase, brain-derived neurotropic factor and vascular endothelial growth factor. Patients will then receive twice-weekly Li-ESWT treatments of 0.2mJ/mm^2 over 3 treatment sites along the dorsal penile shaft, 1500 shocks per treatment (500 shocks per treatment site), for a total of 3000 shocks per week, for 6 weeks of treatment (totally 18,000 shocks). Following Li-ESWT treatments, patients will complete the same validated questionnaires, penile Doppler studies, corporal aspirates and measurement of intracavernosal pressures immediately following the final Li-ESWT treatment, 4-6 weeks following completion of treatment, and again at 3 and 6 months following completion of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male veterans between 40 and 80 years of age
* Known or suspected vasculogenic erectile dysfunction based on clinical history
* In an active sexual relationship with a minimum of 2 sexual attempts per month for at least one month prior to enrollment
* Suffering from ED for at least 6 months
* International Index of Erectile Function - EF domain score between 17-25, Erection Hardness Score score ≥ 1
* Testosterone level between 300-1000ng/dL within one month prior to enrollment
* Hgb A1c ≤ 8% within one month prior to enrollment
* Able to consent to study participation

Exclusion Criteria:

* Erectile dysfunction due to radical prostatectomy, prior pelvic surgery, or radiation therapy to the pelvis within 12 months prior to enrollment.
* Men with known neurogenic or psychogenic ED
* Anatomic malformations of the penis including Peyronie's disease
* Testosterone < 300ng/dL or >1000ng/dL
* Hgb A1c > 8%
* International Normalized Ratio > 2.5, and men on any blood thinners other than 81mg aspirin

Participants will be required to discontinue all erectogenic medications for 1 months prior to initiation of treatment and will not be permitted to use erectogenic medications for the duration of the treatment study.

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants must be men with erectile disfunction.
Enrollment: 25 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Treatment Efficacy | 12 months
  To evaluate the efficacy of the Storz Duolith SD-1 T-top >>ultra<< Li-ESWT device
Treatment Efficacy | 12 months
  To provide data in support of a standardized protocol for the treatment duration for use of this device in treatment of erectile dysfuntion
Treatment Efficacy | 12 months
  To provide data in support of a standardized protocol for the treatment dose for use of this device in treatment of erectile dysfuntion

SECONDARY OUTCOMES:
Measurement of improvements in penile corporal tissues | 12 months
  To evaluate for upregulation of nNOS, eNOS, BDNF and VEGF within penile corporal tissue
Measurement of improvements in penile corporal tissues | 12 months
  To evaluate for improvements in penile blood flow as detectable on penile Doppler and by measurement of intracavernosal pressures
Measurement of improvements in penile corporal tissues | 12 months
  To evaluate for improvements in penile blood flow as detectable by measurement of intracavernosal pressures

CONTACTS AND LOCATIONS:
Locations (1):
- Hunter Holmes McGuire VAMC, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Young SR, Dyson M. The effect of therapeutic ultrasound on angiogenesis. Ultrasound Med Biol. 1990;16(3):261-9. doi: 10.1016/0301-5629(90)90005-w. PMID 1694604
- [Background] Angulo JC, Arance I, de Las Heras MM, Meilan E, Esquinas C, Andres EM. Efficacy of low-intensity shock wave therapy for erectile dysfunction: A systematic review and meta-analysis. Actas Urol Esp. 2017 Oct;41(8):479-490. doi: 10.1016/j.acuro.2016.07.005. Epub 2016 Aug 10. English, Spanish. PMID 27521134
- [Background] Sokolakis I, Dimitriadis F, Psalla D, Karakiulakis G, Kalyvianakis D, Hatzichristou D. Effects of low-intensity shock wave therapy (LiST) on the erectile tissue of naturally aged rats. Int J Impot Res. 2019 May;31(3):162-169. doi: 10.1038/s41443-018-0064-0. Epub 2018 Aug 17. PMID 30120384
- [Background] Liu T, Shindel AW, Lin G, Lue TF. Cellular signaling pathways modulated by low-intensity extracorporeal shock wave therapy. Int J Impot Res. 2019 May;31(3):170-176. doi: 10.1038/s41443-019-0113-3. Epub 2019 Jan 22. PMID 30670837
- [Background] Lin G, Reed-Maldonado AB, Wang B, Lee YC, Zhou J, Lu Z, Wang G, Banie L, Lue TF. In Situ Activation of Penile Progenitor Cells With Low-Intensity Extracorporeal Shockwave Therapy. J Sex Med. 2017 Apr;14(4):493-501. doi: 10.1016/j.jsxm.2017.02.004. Epub 2017 Mar 1. PMID 28258952
- [Background] Vardi Y, Appel B, Jacob G, Massarwi O, Gruenwald I. Can low-intensity extracorporeal shockwave therapy improve erectile function? A 6-month follow-up pilot study in patients with organic erectile dysfunction. Eur Urol. 2010 Aug;58(2):243-8. doi: 10.1016/j.eururo.2010.04.004. Epub 2010 May 6. PMID 20451317
- [Background] Clavijo RI, Kohn TP, Kohn JR, Ramasamy R. Effects of Low-Intensity Extracorporeal Shockwave Therapy on Erectile Dysfunction: A Systematic Review and Meta-Analysis. J Sex Med. 2017 Jan;14(1):27-35. doi: 10.1016/j.jsxm.2016.11.001. Epub 2016 Dec 13. PMID 27986492
- [Background] Man L, Li G. Low-intensity Extracorporeal Shock Wave Therapy for Erectile Dysfunction: A Systematic Review and Meta-analysis. Urology. 2018 Sep;119:97-103. doi: 10.1016/j.urology.2017.09.011. Epub 2017 Sep 27. PMID 28962876
- [Derived] Coffey S, Nguyen V, Matthew AN, Kastelberg BS, Teves ME, Ghatas M, Klausner AP, Smith RP, Krzastek SC. Lack of sustained improvements in erectile function following low-intensity extracorporeal shockwave therapy correlate with decreases in corporal brain-derived neurotropic factor: a pilot study and prospective clinical trial. Sex Med. 2026 Jan 22;13(6):qfaf107. doi: 10.1093/sexmed/qfaf107. eCollection 2025 Dec. PMID 41583708

DOCUMENTS (1):
  • Informed Consent Form (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT04720755/ICF_000.pdf